CLINICAL TRIAL: NCT05090410
Title: Efficacy and Safety of Selective JAK 1 Inhibitor Filgotinib in Active Rheumatoid Arthritis Patients With Inadequate Response to Methotrexate: Comparative Study With Filgotinib and Tocilizumab Examined by Clinical Index as Well as Musculoskeletal Ultrasound Assessment
Brief Title: Efficacy and Safety of Selective JAK 1 Inhibitor Filgotinib in Active Rheumatoid Arthritis Patients With Inadequate Response to Methotrexate
Acronym: TRANSFORM
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Atsushi Kawakami (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor-Investigator, Atsushi Kawakami, Professor, Nagasaki University
Organization: Nagasaki University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRB20_026
Record Dates: First submitted 2021-09-30; First posted 2021-10-22 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Rheumatoid Arthritis; JAK Inhibitor; IL-6 Inhibitor; Musculoskeletal Ultrasound; Biomarker
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — GLPG0634

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Filgotinib monotherapy (Experimental): The administration of filgotinib 200mg/day switched from MTX ± other csDMARDs throughout the study period.
  Interventions: Drug: filgotinib 200mg/day
- Tocilizumab monotherapy (Active Comparator): The administration of subcutaneous tocilizumab 162mg/biweekly switched from MTX ± other csDMARDs throughout the study period.
  Interventions: Drug: subcutaneous tocilizumab 162mg/biweekly

INTERVENTIONS:
Drug: filgotinib 200mg/day — Patients will be randomized in a 1:1 ratio to the administration of filgotinib 200mg/day or subcutaneous tocilizumab 162mg/biweekly switched from MTX ± other csDMARDs throughout the study period.
  Arms: Filgotinib monotherapy
Drug: subcutaneous tocilizumab 162mg/biweekly — Patients will be randomized in a 1:1 ratio to the administration of filgotinib 200mg/day or subcutaneous tocilizumab 162mg/biweekly switched from MTX ± other csDMARDs throughout the study period.
  Arms: Tocilizumab monotherapy

SUMMARY:
The administration of Janus kinase (JAK) inhibitors as well as biological disease-modifying anti-rheumatic drugs has dramatically improved even the clinical outcomes in rheumatoid arthritis (RA) patients with inadequate response to methotrexate (MTX). The dysregulation of JAK-signal transducer and activator of transcription (STAT) pathways via overproduction of cytokines, such as interleukin-6 (IL-6) is involved in the pathogenesis of RA. Filgotinib is a selective JAK1 inhibitor to be approved for use in RA. Filgotinib is effective in suppressing disease activity and preventing the progression of joint destruction due to inhibition of the JAK-STAT pathway. IL-6 inhibitors such as tocilizumab also inhibit the JAK-STAT pathways due to inhibition of IL-6 signaling. We will evaluate whether the effectiveness and safety of filgotinib monotherapy is non-inferior to those of tocilizumab monotherapy in RA patients with inadequate response to MTX.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following requirements to be considered for entry into the study:

  1. ≥20 years old
  2. with the diagnosis of RA based on the ACR/EULAR 2010 RA Classification Criteria
  3. with at least moderate disease activity defined as a DAS28-ESR ≥3.2 at the eligibility evaluation
  4. treated with MTX for ≥8 weeks prior to the providing consent, including 4 weeks or more at the same doses of 8 to 16 mg per week (stable doses of <8 mg per week are allowed only in the presence of intolerance to higher doses)
  5. ability and willingness to provide written informed consent and comply with the requirements of the study protocol

Exclusion Criteria:

* The exclusion criteria are as follows:

  1. concurrent use of a corticosteroid equivalent to >5 mg/day of prednisolone
  2. applicable an item for the contraindication of filgotinib or tocilizumab
  3. a previous use of a JAK inhibitor or IL-6 inhibitor
  4. treatment with a corticosteroid and csDMARD and change of dose within 4 weeks prior to the providing consent
  5. treatment with a biologic DMARD or a biosimilar DMARD (ie, infliximab, biosimilar of infliximab, adalimumab, biosimilar of adalimumab, golimumab, certolizumab pegol or abatacept) within 8 weeks prior to the providing consent
  6. treatment with a TNF inhibitor (ie, etanercept or biosimilar of etanercept) within 4 weeks prior to the providing consent
  7. use of a prohibited drug or therapy, other than the agents noted above, within 4 weeks prior to the providing consent
  8. a complication causing musculoskeletal disorders other than RA (ie, ankylosing spondyloarthritis, reactive arthritis, psoriatic arthritis, crystal-induced arthritis, systemic lupus erythematosus, systemic scleroderma, inflammatory myopathy, or mixed connective tissue disease)
  9. current pregnancy, breastfeeding, or noncompliant with a medically approved contraceptive regimen during and 12 months after the study period
  10. inappropriateness for inclusion in this study as determined by the investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-03-03 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
the proportion of patients who achieve an American College of Rheumatology (ACR) 50 response | at week 12

SECONDARY OUTCOMES:
the proportion of patients who achieve an ACR20 response | at weeks 2, 4, 8, 12, 24, 36 and 52
the proportion of patients who achieve an ACR50 response | at weeks 2, 4, 8, 24, 36 and 52
the proportion of patients who achieve an ACR70 response | at weeks 2, 4, 8, 12, 24, 36 and 52
changes in the clinical disease activity index (CDAI) value | from baseline to weeks 2, 4, 8, 12, 24, 36, and 52
  Higher scores mean a more active of RA.
changes in the simplified disease activity index (SDAI) value | from baseline to weeks 2, 4, 8, 12, 24, 36, and 52
  Higher scores mean a more active RA.
changes in the Disease Activity Score (DAS)28-ESR value | from baseline to weeks 2, 4, 8, 12, 24, 36, and 52
  Higher scores mean a more active RA.
changes in the DAS28-CRP value | from baseline to weeks 2, 4, 8, 12, 24, 36, and 52
  Higher scores mean a more active RA.
changes in the serum levels of biomarkers | from baseline to weeks 2, 4, 12, 24, 36, and 52
  We analyze the serum levels of multiple biomarkers such as cytokines and chemokines.
changes in the total power Doppler (PD) score | from baseline to weeks 4, 12, 24, 36, and 52
  Higher scores mean a more active RA.
changes in the total grayscale (GS) score | from baseline to weeks 4, 12, 24, 36, and 52
  Higher scores mean a more active RA.
changes in the combined PD score | from baseline to weeks 4, 12, 24, 36, and 52
  Higher scores mean a more active RA.
change in van der Heijde-modified total Sharp score (vdH-mTSS) | from baseline to weeks 24 and 52
  Higher scores mean a more joint destruction and deformity.
change in the Health Assessment Questionnaire-Disability Index (HAQ-DI) data | from baseline to weeks 2, 4, 8, 12, 24, 36, and 52
  Higher scores mean a more active RA.
change in the EuroQol 5 Dimensions 5-Level (EQ-5D-5L) data | from baseline to weeks 2, 4, 8, 12, 24, 36, and 52
  Higher scores mean a worse QOL.
change in the Functional Assessment of Chronic Illness-Fatigue (FACIT-F) data | from baseline to weeks 2, 4, 8, 12, 24, 36, and 52
  Higher scores mean a worse fatigue.
changes in the morning stiffness duration | from baseline to weeks 2, 4, 8, 12, 24, 36, and 52
  Higher scores mean a more active RA.
changes in the morning stiffness activity | from baseline to weeks 2, 4, 8, 12, 24, 36, and 52
  We analyze the visual analog scale of morning stiffness activity. Higher scores mean a more active RA.

CONTACTS AND LOCATIONS:
Overall Officials: Atsushi Kawakami, MD, PhD, Principal Investigator — Nagasaki University
Locations (1):
- Nagasaki University Hospital, Nagasaki, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shimizu T, Kawashiri SY, Morimoto S, Kawazoe Y, Kuroda S, Kawasaki R, Ito Y, Kiya R, Sato S, Yamamoto H, Kawakami A. Efficacy and safety of selective JAK 1 inhibitor filgotinib in active rheumatoid arthritis patients with inadequate response to methotrexate: comparative study with filgotinib and tocilizumab examined by clinical index as well as musculoskeletal ultrasound assessment (TRANSFORM study): study protocol for a randomized, open-label, parallel-group, multicenter, and non-inferiority clinical trial. Trials. 2023 Mar 3;24(1):161. doi: 10.1186/s13063-023-07176-5. PMID 36869356